CLINICAL TRIAL: NCT04366843
Title: Impact of Exercises and Chair Massage on Musculoskeletal Pain of Young Musicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Anna Cygańska, Principal Investigator, Master, Józef Piłsudski University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SKE 01-61/2017
Record Dates: First submitted 2020-04-19; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Musculoskeletal Pain
Keywords: musculoskeletal pain; playing related musculoskeletal disorders; physiotherapy
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The chair massage group (Experimental): chair massage 15 min,, 2 x week; measurement before and after each treatment
  Interventions: Other: chair massage
- The exercise program group (Experimental): excercises 15 min., 2 x week; measurement before and after each treatment
  Interventions: Other: the exercise program
- The control group (No Intervention): control 2 measurements, 4 weeks apart

INTERVENTIONS:
Other: chair massage — Chair massage was performed useing only traditional methods of Swedish massage were used, consisting of stroking (smooth, continuous movements to relax and calm the sympathetic nervous system), kneading (consisting of wringing, squeezing muscles, compressing pressure points for the relaxation of soft tissues, i.e. muscles, tendons, fascia), stretching combined with swaying and passive movements of the upper limbs (to mobilize the joints of the upper limbs) and final stroking combined with slapping and shaking percussion, vibration.
  Arms: The chair massage group
Other: the exercise program — The original set of exercises was developed based on the knowledge and clinical experience of the authors of the study and based on EBP (Evidence Based Practice). The program consisted of 14 strengthening and stretching exercises involving the muscles of the trunk and limbs whose main goal was to mobilize the joints and strengthen the weakened muscles and relax overloaded muscle groups.
  Arms: The exercise program group

SUMMARY:
The study is tested the idea of two forms of musculoskeletal pain prophylaxis (chair massage and an original set of exercises) among musicians.

The hypothesis of the study was that massage and exercises could be helpful for musicians to avoid pain conected with playing musical instrument.

ELIGIBILITY:
Inclusion Criteria:

* playing a musical instrument for a minimum of 5 years
* age over 18 years

Exclusion Criteria:

* neurological and oncological diseases
* medical contraindication to undertake physical exercise
* contraindications to perform massage
* lack of consent for participation in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Changes in algometric measurements at 4 weeks | Change between Baseline and post-treatment after 4 weeks
  The algometric measurement concerned the assessment of muscle pressure sensitivity - pain threshold in kg/cm2 made using the Pain Test FPX Algometer (Wagner).

CONTACTS AND LOCATIONS:
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No